CLINICAL TRIAL: NCT06360757
Title: Multi-Center Clinical Performance Evaluation of the NeuMoDx SARS-CoV-2 Assay on the NeuMoDx Molecular Systems
Brief Title: Clinical Evaluation of the NeuMoDx SARS-CoV-2 Assay (COVID-19)
Status: Terminated | Type: Observational
Why Stopped: Discontinuation of product line
Sponsor: QIAGEN Gaithersburg, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: DHF-21-2141-1
Record Dates: First submitted 2024-04-02; First posted 2024-04-11 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2024-04

CONDITIONS: SARS-CoV-2 Acute Respiratory Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Nasopharyngeal swabs in UTM or UVT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: NeuMoDx SARS-CoV-2 Assay — The NeuMoDx™ SARS-CoV-2 Assay is an automated, in vitro nucleic acid amplification test intended for the qualitative detection of SARS-CoV-2 RNA in nasopharyngeal (NP) swabs in transport medium obtained from symptomatic individuals suspected of COVID-19 infection. The NeuMoDx SARS-CoV-2 Assay as performed on the NeuMoDx™ 288 Molecular System and NeuMoDx™ 96 Molecular System incorporates automated RNA extraction to isolate target nucleic acids from the specimen and real-time reverse transcription PCR targeting two conserved regions of the SARS-CoV-2 genome.

SUMMARY:
A multicenter study, using prospectively collected, fresh (Category I) and frozen (Category II), residual/leftover nasopharyngeal (NP) swab in UTM/UVT specimens obtained from symptomatic individuals suspected of COVID-19 infection. This study will evaluate the NeuMoDx SARS-CoV-2 Assay's clinical performance on the NeuMoDx 288 and NeuMoDx 96 Molecular Systems.

ELIGIBILITY:
Inclusion Criteria:

1. Any de-identified NP swab specimen in transport medium from a symptomatic individual suspected of COVID-19 at the time of collection.
2. NP swab specimens obtained using a flexible mini-tip flocked swab and collected into 3mL Copan UTM [Cat. No. 305C] or BD UVT [Cat. No. 220531].
3. Prospective specimens, fresh (Category I) shall be tested within:

   1. (4) hours when held at room temperature, or
   2. (3) days when held at (2 to 8°C), with cold storage starting within (4) hours of collection.
4. Minimum volume of ≥ 2mL.

Exclusion Criteria:

1. Required information unable to be obtained from the associated medical chart.
2. Specimens that remained on-board the NeuMoDx System for > (8) hours prior to processing.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Symptomatic subjects suspected of COVID-19
Sampling Method: Probability Sample
Enrollment: 503 (Actual)
Dates: Start 2024-02-06 (Actual); Primary Completion 2024-07-24 (Actual); Study Completion 2024-07-24 (Actual)

PRIMARY OUTCOMES:
Sensitivity as compared to the comparator method | Through study completion estimated 9 months
  Sensitivity ≥ 95% with a lower bound of the two-sided 95% CI > 90%

SECONDARY OUTCOMES:
Specificity | Through study completion estimated 9 months
  Specificity ≥ 95% with a lower bound of the two-sided 95% CI > 90%

CONTACTS AND LOCATIONS:
Locations (1):
- QIAGEN Gaithersburg, Inc, Manchester, United Kingdom